CLINICAL TRIAL: NCT00107081
Title: A Prospective Multi-Center Study on Pediatric Patients With Fever in Severe Chemotherapy Induced Neutropenia, Including a Randomized Comparison of Outpatient Management and Oral Antimicrobial Therapy Versus Inpatient Management and Intravenous Antimicrobial Therapy in a Subgroup With Low Risk of Adverse Events (Low-Risk Subgroup Study)
Brief Title: Low-risk Fever and Neutropenia in Children With Cancer: Safety and Efficacy of Oral Antibiotics in an Outpatient Setting
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Accrual goal for interventional part not achievable
Sponsor: Swiss Pediatric Oncology Group (Other)
Collaborators: Swiss Cancer League (Other); Bayer (Industry); GlaxoSmithKline (Industry)
Responsible Party: Swiss Pediatric Oncology Group; Roland A Ammann, MD
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPOG 2003 FN; Umbrella Network Trial 2004.3; OCS - 01466-02-2004
Record Dates: First submitted 2005-04-04; First posted 2005-04-05 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Fever; Neutropenia; Cancer
Keywords: children; oral antibiotics; outpatient treatment; fever and neutropenia
MeSH Terms: conditions — Fever; Neutropenia; Neoplasms | interventions — Ciprofloxacin; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (Active Comparator): Continued inpatient i.v. antibiotics
  Interventions: Drug: i.v. antibiotics; Procedure: inpatient management
- Experimental (Experimental): Switch to outpatient p.o. antibiotics
  Interventions: Drug: ciprofloxacin and amoxicillin; Procedure: Outpatient management

INTERVENTIONS:
Drug: ciprofloxacin and amoxicillin
  Arms: Experimental
Procedure: Outpatient management
  Arms: Experimental
Drug: i.v. antibiotics
  Arms: Standard
Procedure: inpatient management
  Arms: Standard

SUMMARY:
The purpose of this study is to determine whether, in children with cancer presenting with fever in severe chemotherapy-induced neutropenia at low risk for medical complications, oral antibiotics in an outpatient setting after an initial phase of intravenous antibiotics and in-hospital observation for 8 to 22 hours, is not inferior as to safety and efficacy compared to continued intravenous antibiotics given in-hospital.

DETAILED DESCRIPTION:
Details on antimicrobial therapy

* At presentation with FN (fever and neutropenia) and during an initial inpatient observation period of 8 to 22 hours, empirical intravenous broad-spectrum antibiotics are given. Type and dosage are chosen by the treating physician.
* Patients randomized to continued intravenous antibiotics continue with these antibiotics.
* Patients randomized to oral antibiotics receive a combination of oral ciprofloxacin (25 to 30 mg/kg/day, top dose 1500 mg/day) plus oral amoxicillin (65 to 80 mg/kg/day, top dose 2250 mg/day), both given in two doses per day.
* In both groups, the study gives guidelines (for certain situations) and rules (for other situations) when to change and when to stop antibiotics.

Details on clinical and laboratory controls

* During antibiotic therapy, patients are seen daily, either as inpatients or as outpatients according to randomization. Complete blood counts are performed at least every second day.
* After stopping antibiotic therapy and until resolution of severe neutropenia (if applicable), patients are seen every other day, with a complete blood count.
* Patients randomized to outpatient management have the possibility to contact at any time of the day (and night) a pediatric oncologist in case of problems, in order to discuss necessity for emergency control and/or rehospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy because of malignancy
* Severe neutropenia (absolute neutrophil count ≤ 0.5x10E9/L)
* Fever (axillary temperature ≥ 38.5°C once or ≥ 38.0°C during ≥ 2 hours)
* Able to swallow oral medication
* Written informed consent from patients and/or parents

Exclusion Criteria:

* Status post myeloablative chemotherapy
* Diagnosis: acute myeloid leukemia, B-cell acute lymphoblastic leukemia, or B-cell Non-Hodgkin lymphoma
* Bone marrow involvement by malignancy ≥ 25%
* Any comorbidity requiring hospitalization: [1] mean arterial blood pressure < 50 mmHg (up to 10 years) / < 60 mmHg (older than 10 years); [2] oxygen saturation < 94% at room air; [3] radiologically defined pneumonia; [4] focal bacterial infection; [5] blood cultures taken at presentation reported positive at reassessment; [6] need for inpatient treatment or observation due to any other reason, as judged by the physician in charge
* Ever shaking chills
* Ever axillary temperature ≥ 39.5°C
* Antibacterial treatment before presentation with fever and neutropenia (except for prevention against Pneumocystis jiroveci [formerly P. carinii] pneumonia)
* Modification or de novo institution of a prophylaxis against P. jiroveci pneumonia
* Modification or de novo institution of a therapy with G-CSF or GM-CSF.
* Allergy to ciprofloxacin and/or amoxicillin
* Serum creatinine level above the upper limit of normal range

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety: No serious medical complication due to infection (death, treatment in ICU [Intensive Care Unit], potentially life-threatening complication) (non-inferiority-design, limit 3.5%)
Efficacy: Response without rehospitalization or changing randomized antibiotics (non-inferiority design, limit 10%)

SECONDARY OUTCOMES:
Improved prediction of low-risk episodes of fever and neutropenia
Description of characteristics of low-risk episodes of fever and neutropenia
Description of characteristics of high-risk episodes of fever and neutropenia (observational study part)

CONTACTS AND LOCATIONS:
Overall Officials: Roland A Ammann, MD, Study Chair — Pediatric Hematology/Oncology, University Children's Hospital, Inselspital, CH-3010 Bern, Switzerland; Christoph Aebi, MD, Study Director — University Children's Hospital, Bern, Switzerland; Maja Beck-Popovic, MD, Principal Investigator — Pediatric Hematology/Oncology, University Children's Hospital, Lausanne, Switzerland; Eveline SJM de Bont, MD, Principal Investigator — Pediatric Hematology/Oncology, University Children's Hospital, Groningen, The Netherlands; Thomas Kuehne, MD, Principal Investigator — Pediatric Hematology/Oncology, University Children's Hospital, Basel, Switzerland; David Nadal, MD, Study Director — University Children's Hospital, Zurich; Felix Niggli, MD, Principal Investigator — Pediatric Hematology/Oncology, University Children's Hospital, Zurich, Switzerland; Arne Simon, MD, Principal Investigator — Pediatric Hematology/Oncology, University Children's Hospital, Bonn, Germany; Nicole Bodmer, MD, Study Director — Pediatric Hematology/Oncology, University Children's Hospital, Zurich, Switzerland; Hulya Ozsahin, MD, Principal Investigator — Pediatric Hematology/Oncology, University Children's Hospital, Geneva, Switzerland
Locations (12):
- Germany (5):
  - Pediatric Hematology/Oncology, University Children's Hospital, Bonn
  - Pediatric Hematology/Oncology, University Children's Hospital, Düsseldorf
  - Pediatric Hematology/Oncology, University Children's Hospital, Freiburg im Breisgau
  - Pediatric Hematology/Oncology, University Children's Hospital von Hauner, Munich
  - Pediatric Hematology/Oncology, University Hospital St. Hedwig, Regensburg
- Pediatric Hematology/Oncology, University Children's Hospital, Groningen, Netherlands
- Switzerland (6):
  - Pediatric Hematology/Oncology, University Children's Hospital, Basel
  - Pediatric Hematology/Oncology, University Children's Hospital, Bern
  - Pediatric Hematology/Oncology, University Children's Hospital, Geneva
  - Pediatric Hematology/Oncology, University Children's Hospital, Lausanne
  - Pediatric Hematology/Oncology, Children's Hospital, Lucerne
  - Pediatric Hematology/Oncology, University Children's Hospital, Zurich

REFERENCES:
- [Background] Ammann RA. SPOG 2003 FN: Risikobeurteilung und risikoadaptierte Behandlung bei Kindern und Jugendlichen mit Fieber in Neutropenie. Paediatrica 16(1): 28-31, 2005.
- [Background] Ammann RA, Simon A, de Bont ES. Low risk episodes of fever and neutropenia in pediatric oncology: Is outpatient oral antibiotic therapy the new gold standard of care? Pediatr Blood Cancer. 2005 Sep;45(3):244-7. doi: 10.1002/pbc.20287. No abstract available. PMID 15747334
- [Result] Ammann RA, Bodmer N, Hirt A, Niggli FK, Nadal D, Simon A, Ozsahin H, Kontny U, Kuhne T, Popovic MB, Luthy AR, Aebi C. Predicting adverse events in children with fever and chemotherapy-induced neutropenia: the prospective multicenter SPOG 2003 FN study. J Clin Oncol. 2010 Apr 20;28(12):2008-14. doi: 10.1200/JCO.2009.25.8988. Epub 2010 Mar 15. PMID 20231680
- [Result] Brack E, Bodmer N, Simon A, Leibundgut K, Kuhne T, Niggli FK, Ammann RA. First-day step-down to oral outpatient treatment versus continued standard treatment in children with cancer and low-risk fever in neutropenia. A randomized controlled trial within the multicenter SPOG 2003 FN study. Pediatr Blood Cancer. 2012 Sep;59(3):423-30. doi: 10.1002/pbc.24076. Epub 2012 Jan 23. PMID 22271702
- [Result] Luthi F, Leibundgut K, Niggli FK, Nadal D, Aebi C, Bodmer N, Ammann RA. Serious medical complications in children with cancer and fever in chemotherapy-induced neutropenia: results of the prospective multicenter SPOG 2003 FN study. Pediatr Blood Cancer. 2012 Jul 15;59(1):90-5. doi: 10.1002/pbc.23277. Epub 2011 Aug 11. PMID 21837771
- [Result] Agyeman P, Aebi C, Hirt A, Niggli FK, Nadal D, Simon A, Ozsahin H, Kontny U, Kuhne T, Beck Popovic M, Leibundgut K, Bodmer N, Ammann RA. Predicting bacteremia in children with cancer and fever in chemotherapy-induced neutropenia: results of the prospective multicenter SPOG 2003 FN study. Pediatr Infect Dis J. 2011 Jul;30(7):e114-9. doi: 10.1097/INF.0b013e318215a290. PMID 21394050
- [Result] Ammann RA, Niggli FK, Leibundgut K, Teuffel O, Bodmer N. Exploring the association of hemoglobin level and adverse events in children with cancer presenting with fever in neutropenia. PLoS One. 2014 Jul 14;9(7):e101696. doi: 10.1371/journal.pone.0101696. eCollection 2014. PMID 25020130
- [Result] Agyeman P, Kontny U, Nadal D, Leibundgut K, Niggli F, Simon A, Kronenberg A, Frei R, Escobar H, Kuhne T, Beck-Popovic M, Bodmer N, Ammann RA. A prospective multicenter study of microbiologically defined infections in pediatric cancer patients with fever and neutropenia: Swiss Pediatric Oncology Group 2003 fever and neutropenia study. Pediatr Infect Dis J. 2014 Sep;33(9):e219-25. doi: 10.1097/INF.0000000000000326. PMID 24618935
- [Result] Ammann RA, Bodmer N, Simon A, Agyeman P, Leibundgut K, Schlapbach LJ, Niggli FK. Serum Concentrations of Mannan-Binding Lectin (MBL) and MBL-Associated Serine Protease-2 and the Risk of Adverse Events in Pediatric Patients With Cancer and Fever in Neutropenia. J Pediatric Infect Dis Soc. 2013 Jun;2(2):155-61. doi: 10.1093/jpids/pit005. Epub 2013 Feb 13. PMID 26619462
- See also: The Swiss Pediatric Oncology Group (SPOG) was the sponsor of this study. — http://www.spog.ch